CLINICAL TRIAL: NCT03830983
Title: Atrial Cardiomyopathy in Patients With Stroke of Undetected Mechanism
Status: Completed | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Rigshospitalet, Denmark (Other); Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Ahmad Sajadieh, MD, DMSc, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: 18055313
Record Dates: First submitted 2019-01-29; First posted 2019-02-05 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Stroke
Keywords: Cardioembolic stroke; Cardiac MRI; Heart disease; Vascular disease
MeSH Terms: conditions — Stroke; Embolic Stroke; Heart Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For use in future studies of biomarkers and genes we will collect 2 samples of plasma and 1 sample of full blood. Only patient who give informed consent will have these samples collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stroke of likely cardioembolic cause or undetected mechanism: Lesions in at least one territory on MRI & absence of significant large vessel disease defined as stenosis of cerebral or pre-cerebral vessels >50% in arteries supplying the ischemic area(s) & absence of severe small vessel disease including micro-bleeds on Patients with central retinal artery occlusion documented by perimeter and absence of significant large vessel disease defined as stenosis of cerebral or pre-cerebral vessels >50% & absence of severe small vessel disease including micro-bleeds on MRI are included independent of acute MRI findings.
- Atherosclerotic stroke: Large vessel stroke: Acute lesions in one vascular territory on MRI, significant large vessel disease defined as stenosis of cerebral or pre-cerebral vessels >50% leading to the infarcted territory & absence of severe small vessel disease including micro-bleeds on MRI Small Vessel stroke: MRI documenting lacunar infarction, absence of significant large vessel disease defined as stenosis of cerebral or pre-cerebral vessels >50% and presence of severe small vessel disease possibly including micro bleeds.
- Controls: Age and sex matched healthy controls with no history of stroke or AF.

SUMMARY:
The goal of this study is to evaluate left atrial structural and functional abnormalities in stroke of undetected mechanism and atherosclerotic stroke with cardiac MRI.

DETAILED DESCRIPTION:
Aims and objectives:

The goal of this study is to evaluate left atrial structural and functional abnormalities in patients with stroke of likely cardio-embolic origin compared with healthy age and sex matches controls and patients with atherosclerotic stroke using cardiac MRI.

Background:

Despite standard work up for the etiology of ischemic stroke, about 30% of the cases remain unexplained. It is increasingly accepted that these unexplained cases arise from disease outside of the brain. Paroxysmal AF (Atrial fibrillation) may often be suspected as the source but fewer than one third of patients with stroke of undetermined source manifest AF in any form even after 3 years of continuous heart rhythm monitoring. Emerging evidence suggest that atrial functional and structural abnormalities may convey a comparable risk of stroke in which AF is only one of several features. These abnormalities have been termed "atrial cardiomyopathy" and may be an efficient and practical approach to identify patients at high risk of AF and ischemic stroke.

Methods and materials:

Cross sectional and prospective cohort study with 3 different groups: 50 patients with stroke of undetected mechanism, 50 patients with atherosclerotic stroke (large or small vessel disease) admitted to the University Hospital of Bispebjerg and Frederiksberg and 50 sex and age matched controls with no history of stroke or AF from the Copenhagen City Heart Study (ØBUS) will be included during a 2 year-period. The study will measure atrial structural abnormalities using cardiac magnetic resonance imaging (MRI) and atrial functional abnormalities by cardiac MRI and echocardiography. A 1 year follow up will examine the incidence of silent brain infarction with MRI and incidence of stroke, atrial fibrillation, acute myocardial infarction and cardiovascular death. Secondary endpoints are to examine the association of functional and structural changes found by MRI with echocardiography, rhythm abnormalities and biomarkers with the purpose of finding clinical easily applicable methods to diagnose atrial cardiomyopathy.

Expected outcome and perspectives:

The investigators hypothesize that patients with stroke of likely cardio-embolic origin have significantly more atrial fibrotic degeneration and reduced atrial emptying function than patients with atherosclerotic stroke and the control subjects. The investigators expect a higher incidence of silent brain infarction in the group with stroke of likely cardio-embolic origin. With atrial cardiomyopathy investigated thoroughly in patients with stroke of likely cardio-embolic origin the future work-up and treatment strategies could be more efficient and may thus improve the prognosis in terms of mortality and disability for a considerable number of patients.

ELIGIBILITY:
Inclusion Criteria (Patients):

1. Stroke of likely cardioembolic cause or of undetected mechanism:

   Lesions in at least one territory on MRI & absence of significant large vessel disease defined as stenosis of cerebral or pre-cerebral vessels >50% in arteries supplying the ischemic area(s) & absence of severe small vessel disease including micro-bleeds on MRI.

   Patients with central retinal artery occlusion documented by perimeter and absence of significant large vessel disease defined as stenosis of cerebral or pre-cerebral vessels >50% & absence of severe small vessel disease including micro-bleeds on MRI are included independent of acute MRI findings.
2. Large or small vessel stroke (atherosclerotic stroke):

   Large vessel stroke: Acute lesions in one vascular territory on MRI, significant large vessel disease defined as stenosis of cerebral or pre-cerebral vessels >50% leading to the infarcted territory & absence of severe small vessel disease including micro-bleeds on MRI Small Vessel stroke: MRI documenting lacunar infarction, absence of significant large vessel disease defined as stenosis of cerebral or pre-cerebral vessels >50% and presence of severe small vessel disease possibly including micro bleeds.
3. Ischemic stroke within 30 days prior to inclusion
4. Age > 18 years
5. Life expectancy of at least one year
6. Informed consent

   * Stenosis: % defined by Ultrasound
   * Small vessel disease: defined according to STRIVE criteria

Inclusion Criteria (Controls)

1. Age and sex matched healthy controls. Matched with the group with stroke of likely cardioembolic stroke.

Exclusion Criteria (Patients):

1. Prior AF or AF >30 sec on at least 6 hours of monitoring during hospitalization.
2. Other major cardio-embolic risk sources assumed as cause of stroke (e.g. endocarditis, myocardial infarction within last 4 weeks, prosthetic cardiac valve)
3. Contraindications to MRI (Including eGFR<30 or other contraindications for the contrast agent used during Cardiac MRI)
4. Assumed unable to participate in the study by investigator (including but not restricted to psychiatric condition, dementia)

Exclusion Criteria (Controls):

1. History of stroke or AF
2. Contraindications to MRI (Including eGFR<30 mL/min/1.73 m2 or other contraindications for the contrast agent used during Cardiac MRI)
3. Assumed unable to participate in the study by the investigator (For the same reasons listed above)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are selected amongst individuals admitted with acute stroke to Bispebjerg University Hospital. Healthy controls will be invited from the the Copenhagen City Heart Study (ØBUS).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Extent of the fibrosis in the Left Atrium (LA) | Within 12 weeks from index event
  Measured with gadolinium enhanced cardiac MRI
Left Atrial Emptying Function (LAEF) | Within 12 weeks from index event
  Measured with gadolinium enhanced cardiac MRI

SECONDARY OUTCOMES:
Observational study: Incidence of silent brain infarctions | Between 1-2 years from index event
  Incidence of silent brain infarctions assessed by follow-up MR-cerebrum (Only in patients)
Left atrial volume | Within 12 weeks from index event
  Assessed by cardiac MRI
Left atrial appendage morphology | Within 8 weeks from index event
  Assessed by cardiac MRI
Left atrium volume | Within 12 weeks from index event
  2D and 3D left atrial volume assessed by transthoracic echocardiography
Left atrium ejection fraction (LAEF) | Within 12 weeks from index event
  Assessed by transthoracic echocardiography
Speckle tracking of LA | Within 12 weeks from index event
  Assessed by transthoracic echocardiography
Atrial rhythm abnormalities: Number of premature atrial contractions (PAC) per hour. Number and length of runs of PAC | Within 4 weeks from index event
  Assessed by 48-hours Holter monitoring
Heart rate variability (HRV) | Within 4 weeks from index event
  Time domain variables (meanNN, SDNN, SDANN, SDNNidx, RMSSD, pNN50)
Thrombophilia biomarkers | Within 12 weeks from index event
  Assessment of hypercoagulability
Cardiac specific biomarkers | Within 12 weeks from index event
  Atrial Natriuretic Peptide, pro NT-Brain Natriuretic Peptide, High Sensitive Troponins.
Inflammatory biomarkers | Within 12 weeks from index event
  High Sensitive CRP, Interleukins: IL1, IL1b, IL6, IL18
Fibrosis related markers | Within 12 weeks from index event
  Collagen type I and III

OTHER OUTCOMES:
Observational study: Assessing incidence of stroke, acute myocardial infarction, atrial fibrillation and cardiovascular-death | 1 year from last included patient
  Follow up in patient records

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Sajadieh, MD, DMSc, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be made available to other research groups upon reasonable request.

REFERENCES:
- [Derived] Larsen BS, Aplin M, Host N, Dominguez H, Christensen H, Christensen LM, Havsteen I, Prescott E, Jensen GB, Vejlstrup N, Bertelsen L, Sajadieh A. Atrial cardiomyopathy in patients with ischaemic stroke: a cross-sectional and prospective cohort study-the COAST study. BMJ Open. 2022 May 11;12(5):e061018. doi: 10.1136/bmjopen-2022-061018. PMID 35545392